CLINICAL TRIAL: NCT03708484
Title: Effect of Aerobic Interval Training Versus Resistance Interval Training on Ejection Fraction in Post Stable Myocardial Infarction Patients
Brief Title: Aerobic Interval Training v/s Resistance Interval Training On Ejection Fraction In Stable Post MI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RiphahIU Hania Farheen
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Myocardial Infarction
Keywords: Aerobic Interval training; Ejection Fraction; Myocardial Infarction; Resistive Interval Training
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Interval Training (Active Comparator): Aerobic Interval Training is active comparator
  Interventions: Other: Aerobic Interval Training
- Aerobic + Resistive Interval Training (Experimental): Aerobic + Resistive Interval Training is experimental
  Interventions: Other: Aerobic + Resistive Interval Training

INTERVENTIONS:
Other: Aerobic Interval Training — Aerobic Interval Training Patients in this group will perform 6 minutes of cycling followed by 3 minutes of pause and again 6 minutes of cycling followed by 3 minutes of pause and finally 6 minutes of treadmill followed by 3 minutes of rest.
  both groups will perform cool down exercises that include again breathing exercises, stretching and active exercises.
  Arms: Aerobic Interval Training
Other: Aerobic + Resistive Interval Training — Aerobic + Resistive Interval Training Patients in this group; first set will perform 3 minute of cycling ,1 set of hand grippers 1.5 to 2.5 lbs (10 to 12 reps) and 1 set of biceps resistive exercises 1 Kg to 3 kg (10 to 12 reps) followed by 3minute of pause. In second set patient will perform 3 minutes of stationary cycling , 1 set of quadriceps resistive exercises 1 to 3 Kg (10 to 12 reps) again followed by 3 minutes of pause and in third set patient will perform 3 minutes of treadmill walk at 1.5 to 4 speed, and 1 set of standing ankle pumps (10 to 12 reps).
  both groups will perform cool down exercises that include again breathing exercises, stretching and active exercises.
  Arms: Aerobic + Resistive Interval Training

SUMMARY:
Randomized controlled trial (single blinded) study was conducted on 26 stable Post MI patients according to inclusion and exclusion criteria aged 35 to 65 years. Study was conducted in Rawalpindi Institute of cardiology and Pakistan Railway Hospital from July 2016 ---- December 2016.Participants was randomly allocated in control or experimental group by lottery Method. Informed consent was signed by each participant prior to enrolment. Patients in both group received standard treatment that is Aerobic Interval training whereas patients in interventional group received additional Resistance training. Post echocardiography and lipid profile was done to assess the effect of intervention on ejection fraction, cholesterol and triglycerides. The standard questionnaire Mac New QLMI was used to assess quality of life. The data was analyzed on SPSS 21

DETAILED DESCRIPTION:
It is already established worldwide that myocardial infarction is one of the leading cause of morbidity and mortality. According to WHO (2008), cardiovascular diseases account for one third of annual deaths. Globally over 17 Million deaths occur each year due to coronary artery diseases. In United States of America, CAD has affected more than 13 million of the population in the year 2003 including almost 860, 000 people with acute MI, whereas 480,000 people lost their lives due to CAD. The prevalence of coronary artery disease in a population can be estimated by incidence of MI in that population.

However, in the past few decades cardiovascular disease rates have considerably decreased in high income countries, but on the other hand have increased in low and middle income countries with 80 percent of global burden of disease in these countries. Global strategy is therefore required to educate about the importance of risk factors in prevention of disease, disability and death and improving clinical outcomes to prevent recurrent event.

Myocardial infarction can be a tragic and a disastrous event leading to sudden death or it can also be a minor event which may even go undetected. Patients who once have MI, always have a chance to get it over and over again.The incidence rate of MI increases with age, particularly after 45 years in men and after 55 years in women. Recurrent infarctions were found more frequent in women than men. First infarction sometimes goes unrecognized but recurrent infarctions were almost always easily recognized.

One of the major complications affecting patient lifestyle after CABG is depression. It affects almost 30 to 40% of the patients undergoing surgery. Evidence also suggests that depression after surgery was more common among those patients who were depressed prior to surgery too. Depression along with anxiety can increase the risk of mortality and morbidity independently without involving any medical cause. Depression and anxiety although do not have that much effect on neuropsychological dysfunction but the risk of disorientation and confusion leading to delirium is increased. Therefore, psychological counseling of patients should be done before surgery to reduce the risk of depression following surgery in order to improve overall quality of life of patient.

Cardiac rehabilitation after discharge from hospital is phase 2 or outpatient cardiac rehabilitation. Phase 2 Rehabilitation is under complete supervision of cardiologist along with physiotherapist, exercise therapist and nurse. Blood pressure and heart rate are monitored at rest during and after exercise session along with ECG monitoring. Phase 2 includes aerobic training that includes treadmill and cycling together with resistance training that can be with hand grippers and weights. Recommended guidelines of exercises are followed which varies according to patients condition and response. Total exercise session is of 50- 60 minutes, prescribed weeks of exercise in low, moderate and high risk patients is of 4, 6 and 8 weeks respectively. Patients are also educated for modification of risk factors, nutritional counseling, weight control and stress management. After competition of phase 2, patients are encouraged to enter maintenance phase that is phase 3.

For an exercise prescription plan, heart rate and metabolic equivalent [1 MET=3.5mL 02/kg/min] is set at 50-80% of the peak during exercise stress testing, or heart rate of 10 or >10 bpm below the ischemic ECG (^0.1 mV), or anginal threshold. In patients who are not tested by exercise testing, 20- 30 beats above their resting heart rate is considered to be the target heart rate. For intensity guide along with heart rate RPE (6-20 scale) is also used. In early stage of phase 2 rehab 11- 13 is considered upper limit for training. However for phase 3, 12- 14 is upper limit and considered safe.

The exercise plan should be individualized according to patient capacity, risk factors and co-morbidities. The universal guidelines of exercise should be followed. Exercise should be started with warm up, followed by prescribed exercise like aerobic and interval training and ending session with cooling to stable patient. Continuous monitoring of vitals is necessary in MI patients during exercise. The progression of exercise is increasing the intensity of exercise with following weeks according to patient's capacity.

In athletes to gain aerobic and anaerobic health, interval training at 75% VO2 max is usually beneficial than traditional continuous training. More recently interval training is introduced. Many studies are done on efficacy and safety of interval training in coronary artery patients but data is still lacking. Furthermore studies are required with larger samples for safe dosage and prescription of interval training in cardiac patients.

Aerobic interval training was found to be more effective than conservative continuous training at moderate intensity in reversing myocardial remodeling post MI as it increases myocardial contractility which has positive effect on ejection fraction, stroke volume and ejection velocity.

One of the studies done by Ehsani in 2007 has found that two of the major factors in remodeling post MI that is resting diastolic diameter and volume of LV decreased in both training groups. While other three factors responsible for increasing heart contractility like ejection fraction, stroke volume and cardiac output only increased in interval training group. In comparison to aerobic training, interval training has no safety hazard. The improvement of muscle strength, body strength and overall cardiac fitness is even better than traditional aerobic training.

Previously only aerobic training was considered safe in coronary artery diseases patients. Resistance training beneficial effects in heart diseases were not established previously considering that resistance training can be harmful as they can cause further ischemia or unlikely events like arrhythmias, especially isometrics were not considered safe in MI patients as many studies reported that they can cause life threatening events like arrhythmias. Previously one of the other reasons for contraindication of resistance training was increased after load causing adverse effect on left ventricular function but recently studies had confirmed that resistance exercise can be an effective mean of therapy in cardiac patients as it has no negative effect on left ventricular function.

After acute MI, resistance exercises are absolutely contraindicated for 2-3 weeks .They can be started slowly after 3 weeks with very low weight of 1-2 lbs with a recommended safe dose of 10-15 reps performed on alternating days and a maximum RPE of 12 to 13. Intensity increases according to individual patient. After 6 weeks of myocardial infarction have passed, weight machines and barbells can be used as a part of resistance training program. Plan of resistance exercises in cardiac patients should be individualized to each patient according to their CV status co-morbidities and degree of LV dysfunction. One of the recommended guidelines for resistance exercises is 2-3 days a week with moderate to high intensity for almost 3-6 months.

Comparison of heart rate and systolic blood pressure changes in cardiac patients during aerobic and resistance training was done. The study showed that peak heart rate was 12% greater than target heart rate during aerobics whereas on other hand it was 12% less than target heart rate during resistance training. Blood pressure monitoring at end of both trainings showed increase in systolic BP was slightly greater than aerobic training.

Many factors contribute to development of atherosclerosis. The role of lipid profile in development of coronary artery diseases in past few decades has been well established The benefits of physical activities are various one of the positive effect seen is on lipid profile with increase in HDL and decrease in total cholesterol and triglycerides alone or together with dietary modifications which are essential component. Aerobic training at moderate to high intensity variably cause an improvement in lipid profile Studies have shown that reduction in triglycerides were seen more in males in comparison to females.

Exercise at low training can also decrease triglycerides from 8 to 20 mgdl with minimum exercise of 24 to 32 km/week and caloric expenditure of 1200 to 2200 Kcal/week. Exercise that reaches this minimum range can produce positive lipid changes.

Combined Strength and aerobic training of 8 months can make positive biochemical and muscular accommodation on total cholesterol triglycerides as well as on HDL. However the changes are reversed with three months of detraining concluding that exercise should be integral part of life as it plays vital role to prevent coronary artery disease.

Exercise training as an integral component of cardiac rehabilitation is intended to restore health and fitness to patients suffering from heart diseases. It has a favorable effect on numerous cardiac and health related outcomes. Left ventricle impairment is a substantial prognostic indicator of mortality. Particularly for coronary heart disease patients, one of the clinical predictors of long-term prognosis is left ventricular ejection fraction (LVEF) which is a marker of myocardial contractility. Ejection fraction is the quantity of blood pumped by the left ventricle of heart per minute into the aorta which is the largest artery in the body. LVEF ≥ 50% is deemed normal, also termed as preserved ejection fraction. Ejection fraction falls considerably after MI and cardiac surgeries such as CABG and valve replacement surgeries. In these patients who undergo heart surgery, phase I cardiac rehabilitation plays a significant role in improving the hemodynamic variables such as ejection fraction.

The effectiveness of phase I cardiac rehabilitation in cardiac surgeries is well-established. But regarding phase II, there is a paucity of accurate data on the effectiveness of various types of exercise training on LVEF in coronary artery disease patients. Most of the studies conducted previously, have explored the impact of exercise on ejection fraction in heart failure patients, whereas methodological disparities are evident in the ones conducted on CAD patients. Therefore, attention is being focused towards this aspect for the past few years. It was found that a 12 weeks structured, individually adapted exercise plan, if started early i.e. within one month after discharge, could considerably improve left ventricle function in terms of LVEF in CAD patients. After consultation with the rehab specialist, the exercise plan could also be carried out at home, if access to a clinical setting is difficult. As impaired LV systolic function is an absolute predictor of mortality in myocardial infarction, hence utilizing cardiac rehab and secondary prevention for improving ejection fraction would result in better survival chances.

My current study aim was to evaluate and find out whether the combination of Resistance interval training and Aerobic interval training is more effective than Aerobic interval training alone in improving EF in Post Stable MI patients. This study will add to literature and fill the gap as most studies previously done was on Aerobic interval training in CAD . More over no study has individually focused on post MI patients without surgical interventions. Furthermore No research up to date has compared Aerobic interval training with Resistance interval training in improving EF after MI.

ELIGIBILITY:
Inclusion Criteria:

* Patient who experienced just 1 episode of MI
* Stable post MI patients after 6 weeks of MI episode
* Patient who remained asymptomatic for first 3 minutes of ETT

Exclusion Criteria:

* Poor LV ejection fraction below 35 % was excluded
* Lung diseases ( lung function test moderate and severe intensity )
* Unstable MI patients
* Those who had undergone any cardiac surgery
* Patients with Post MI Arrhythmias were excluded

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-25 (Actual)

PRIMARY OUTCOMES:
Ejection Fraction | 6 weeks
  Change from baseline Ejection fraction

SECONDARY OUTCOMES:
MACNEW QLMI | 6 weeks
  change from Baseline MACNEW QLMI is a self-administered heart disease-specific health-related quality of life [HRQL] instrument. The MacNew is designed to evaluate the impact of treatment, including cardiac rehabilitation, and has been shown to be valid, reliable and responsive, is simple to administer and well-accepted by patients, and normative data are available for patients with myocardial infarction, angina pectoris, and heart failure.
  The Mac New has total of 27 items with three major categories. 14 item emotional function Domain scale, 13 item physical limitations domain scale and 13 item social function domain scale. Scoring of Mac New is simple and easy. Minimum score is 1 that is poor and maximum is 7 that are high score. Missing responses are not scored. Each category is calculated as average of responses in that category.
Lipid profile | 6 weeks
  change from baseline (Lipid profile)

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PHD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction. Universal definition of myocardial infarction. J Am Coll Cardiol. 2007 Nov 27;50(22):2173-95. doi: 10.1016/j.jacc.2007.09.011. No abstract available. PMID 18036459
- [Background] Cornish AK, Broadbent S, Cheema BS. Interval training for patients with coronary artery disease: a systematic review. Eur J Appl Physiol. 2011 Apr;111(4):579-89. doi: 10.1007/s00421-010-1682-5. Epub 2010 Oct 23. PMID 20972578
- [Background] Suaya JA, Shepard DS, Normand SL, Ades PA, Prottas J, Stason WB. Use of cardiac rehabilitation by Medicare beneficiaries after myocardial infarction or coronary bypass surgery. Circulation. 2007 Oct 9;116(15):1653-62. doi: 10.1161/CIRCULATIONAHA.107.701466. Epub 2007 Sep 24. PMID 17893274
- [Background] Kannel WB, Abbott RD. Incidence and prognosis of unrecognized myocardial infarction. An update on the Framingham study. N Engl J Med. 1984 Nov 1;311(18):1144-7. doi: 10.1056/NEJM198411013111802. PMID 6482932
- [Background] Alpert JS, Thygesen K, Antman E, Bassand JP. Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. J Am Coll Cardiol. 2000 Sep;36(3):959-69. doi: 10.1016/s0735-1097(00)00804-4. PMID 10987628
- [Background] Tully PJ, Baker RA. Depression, anxiety, and cardiac morbidity outcomes after coronary artery bypass surgery: a contemporary and practical review. J Geriatr Cardiol. 2012 Jun;9(2):197-208. doi: 10.3724/SP.J.1263.2011.12221. PMID 22916068
- [Background] Wenger NK. Current status of cardiac rehabilitation. J Am Coll Cardiol. 2008 Apr 29;51(17):1619-31. doi: 10.1016/j.jacc.2008.01.030. PMID 18436113
- [Background] Taylor RS, Brown A, Ebrahim S, Jolliffe J, Noorani H, Rees K, Skidmore B, Stone JA, Thompson DR, Oldridge N. Exercise-based rehabilitation for patients with coronary heart disease: systematic review and meta-analysis of randomized controlled trials. Am J Med. 2004 May 15;116(10):682-92. doi: 10.1016/j.amjmed.2004.01.009. PMID 15121495
- [Background] Williams MA, Ades PA, Hamm LF, Keteyian SJ, LaFontaine TP, Roitman JL, Squires RW. Clinical evidence for a health benefit from cardiac rehabilitation: an update. Am Heart J. 2006 Nov;152(5):835-41. doi: 10.1016/j.ahj.2006.05.015. PMID 17070142
- [Background] Gielen S, Laughlin MH, O'Conner C, Duncker DJ. Exercise training in patients with heart disease: review of beneficial effects and clinical recommendations. Prog Cardiovasc Dis. 2015 Jan-Feb;57(4):347-55. doi: 10.1016/j.pcad.2014.10.001. Epub 2014 Oct 22. PMID 25459973
- [Background] Blanchard CM, Courneya KS, Rodgers WM, Fraser SN, Murray TC, Daub B, Black B. Is the theory of planned behavior a useful framework for understanding exercise adherence during phase II cardiac rehabilitation? J Cardiopulm Rehabil. 2003 Jan-Feb;23(1):29-39. doi: 10.1097/00008483-200301000-00007. PMID 12576910
- [Background] Franklin BA, Bonzheim K, Gordon S, Timmis GC. Safety of medically supervised outpatient cardiac rehabilitation exercise therapy: a 16-year follow-up. Chest. 1998 Sep;114(3):902-6. doi: 10.1378/chest.114.3.902. No abstract available. PMID 9743182
- [Background] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726
- [Background] Molmen-Hansen HE, Stolen T, Tjonna AE, Aamot IL, Ekeberg IS, Tyldum GA, Wisloff U, Ingul CB, Stoylen A. Aerobic interval training reduces blood pressure and improves myocardial function in hypertensive patients. Eur J Prev Cardiol. 2012 Apr;19(2):151-60. doi: 10.1177/1741826711400512. Epub 2011 Mar 4. PMID 21450580
- [Background] Kemi OJ, Wisloff U. High-intensity aerobic exercise training improves the heart in health and disease. J Cardiopulm Rehabil Prev. 2010 Jan-Feb;30(1):2-11. doi: 10.1097/HCR.0b013e3181c56b89. PMID 20040880
- [Background] Karlsdottir AE, Foster C, Porcari JP, Palmer-McLean K, White-Kube R, Backes RC. Hemodynamic responses during aerobic and resistance exercise. J Cardiopulm Rehabil. 2002 May-Jun;22(3):170-7. doi: 10.1097/00008483-200205000-00008. PMID 12042685
- [Background] Pollock ML, Franklin BA, Balady GJ, Chaitman BL, Fleg JL, Fletcher B, Limacher M, Pina IL, Stein RA, Williams M, Bazzarre T. AHA Science Advisory. Resistance exercise in individuals with and without cardiovascular disease: benefits, rationale, safety, and prescription: An advisory from the Committee on Exercise, Rehabilitation, and Prevention, Council on Clinical Cardiology, American Heart Association; Position paper endorsed by the American College of Sports Medicine. Circulation. 2000 Feb 22;101(7):828-33. doi: 10.1161/01.cir.101.7.828. No abstract available. PMID 10683360
- [Background] Cornelissen VA, Fagard RH, Coeckelberghs E, Vanhees L. Impact of resistance training on blood pressure and other cardiovascular risk factors: a meta-analysis of randomized, controlled trials. Hypertension. 2011 Nov;58(5):950-8. doi: 10.1161/HYPERTENSIONAHA.111.177071. Epub 2011 Sep 6. PMID 21896934
- [Background] Leon AS, Sanchez OA. Response of blood lipids to exercise training alone or combined with dietary intervention. Med Sci Sports Exerc. 2001 Jun;33(6 Suppl):S502-15; discussion S528-9. doi: 10.1097/00005768-200106001-00021. PMID 11427777
- [Background] Tokmakidis SP, Volaklis KA. Training and detraining effects of a combined-strength and aerobic exercise program on blood lipids in patients with coronary artery disease. J Cardiopulm Rehabil. 2003 May-Jun;23(3):193-200. doi: 10.1097/00008483-200305000-00006. PMID 12782903
- [Background] White HD, Norris RM, Brown MA, Brandt PW, Whitlock RM, Wild CJ. Left ventricular end-systolic volume as the major determinant of survival after recovery from myocardial infarction. Circulation. 1987 Jul;76(1):44-51. doi: 10.1161/01.cir.76.1.44. PMID 3594774
- [Background] Meta-analysis Global Group in Chronic Heart Failure (MAGGIC). The survival of patients with heart failure with preserved or reduced left ventricular ejection fraction: an individual patient data meta-analysis. Eur Heart J. 2012 Jul;33(14):1750-7. doi: 10.1093/eurheartj/ehr254. Epub 2011 Aug 6. PMID 21821849
- [Background] Haddadzadeh MH, Maiya AG, Padmakumar R, Shad B, Mirbolouk F. Effect of exercise-based cardiac rehabilitation on ejection fraction in coronary artery disease patients: a randomized controlled trial. Heart Views. 2011 Apr;12(2):51-7. doi: 10.4103/1995-705X.86013. PMID 22121461
- [Background] Pierson LM, Herbert WG, Norton HJ, Kiebzak GM, Griffith P, Fedor JM, Ramp WK, Cook JW. Effects of combined aerobic and resistance training versus aerobic training alone in cardiac rehabilitation. J Cardiopulm Rehabil. 2001 Mar-Apr;21(2):101-10. doi: 10.1097/00008483-200103000-00007. PMID 11314283
- [Background] Kang K, Gholizadeh L, Inglis SC, Han HR. Interventions that improve health-related quality of life in patients with myocardial infarction. Qual Life Res. 2016 Nov;25(11):2725-2737. doi: 10.1007/s11136-016-1401-8. Epub 2016 Sep 3. PMID 27592108

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT03708484/Prot_SAP_002.pdf
  • Informed Consent Form (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT03708484/ICF_003.pdf